CLINICAL TRIAL: NCT00840190
Title: An Open Label, Multicenter Phase I Study Of Selective Cyclin Dependent Kinase Inhibitor P1446A-05 In Subjects With Advanced Refractory Malignancies
Brief Title: A Study Of Selective Cyclin Dependent Kinase Inhibitor P1446A-05 In Subjects With Advanced Refractory Malignancies
Acronym: Serenity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1446A-05/19/08
Record Dates: First submitted 2009-02-03; First posted 2009-02-10 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Solid Tumor; Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P1446A-05 (Experimental)
  Interventions: Drug: P1446A-05

INTERVENTIONS:
Drug: P1446A-05 — P1446A-05 available as 25mg,50mg,100mg capsule. Subjects will be enrolled at at different dose levels of P1446A-05 to be taken once a day for 14 days followed by 7 days rest.This constitutes one cycle of P1446A-05. Four such cycles will be administered.

SUMMARY:
This is a phase I open label study to evaluate safety and efficacy of P1446A-05 in subjects with advanced refractory malignancies. Subjects of solid tumors or hematologic malignancies will be included. This is a dose escalation study following an accelerated titration design. It is expected that around 50 subjects would be enrolled in the study.Safety assessment will be conducted on the basis of vital signs, physical examination and laboratory investigations undertaken at regular intervals as per the schedule.

DETAILED DESCRIPTION:
This is a phase I open label study to evaluate safety and efficacy of P1446A-05 in subjects with advanced refractory malignancies. Subjects of solid tumors or hematologic malignancies will be included as per selection criteria. Starting dose for P1446A-05 in this study is 75 mg orally once daily for 14 days followed by 7 days rest. This constitutes one cycle for P1446A-05.Three patients will be enrolled in first cohort at this starting dose of P1446A-05. If this dose is well tolerated then dose escalation will be undertaken for subsequent cohorts as per accelerated titration design as described in protocol till maximum tolerated dose(MTD) for P1446A-05 is determined. The MTD will be the recommended phase 2 dose. 10 additional patients might be enrolled at this MTD to further evaluate safety and efficacy. It is expected that around 50 subjects would be enrolled in the study.Safety assessment will be conducted on the basis of vital signs, physical examination and laboratory investigations undertaken at regular intervals as per the schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically and/ or cytologically confirmed solid malignant tumor or hematologic malignancy that is refractory to currently available treatment or for which no standard treatment exists
2. Subjects of either sex and more than or equal to 18 years of age
3. ECOG (Eastern Cooperative Oncology Group) performance status less than or equal to 2
4. Subjects with life expectancy of at least 4 months
5. Hemoglobin greater than or equal to 8 g/dl
6. Absolute neutrophil count greater than or equal to 1000/mm3
7. Platelet count greater than or equal to 50,000/ mm3
8. Total bilirubin less than or equal to 1.5 X institutional upper limit of normal (ULN)
9. AST/ALT less than or equal to 3 X institutional upper limit of normal (ULN)
10. Creatinine less than or equal to 1.5 X institutional upper limit of normal (ULN)
11. Ability to understand and willingness to sign a written informed consent document.

Exclusion criteria

1. Subjects who have received radiotherapy, chemotherapy or biologic/targeted anticancer agents within 4 weeks prior to day 1 of study drug administration (6 weeks for nitrosoureas or mitomycin C) or have not recovered completely from adverse effects of any prior radiotherapy, chemotherapy or biologic/targeted agents
2. Subjects who have received autologous or allogeneic bone marrow transplant within 6 months of day 1 of study drug administration
3. Subjects with known brain metastases at the time of screening
4. Subjects who had received any other investigational drug within 1 month or within five half-lives of the other investigational agent, whichever is longer prior to day 1 of study drug administration or who have not completely recovered from adverse effects of the investigational agent received prior to this period.
5. History of allergic reactions attributed to compounds of similar chemical structure to P1446A-05.
6. Subjects on immunosuppressive therapy.
7. History of unstable angina or myocardial infarction or stroke within previous 6 months.
8. Subjects with uncontrolled inter-current illness including, but not limited to active infection, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Subjects known to be suffering from infection with HIV, Tuberculosis, Hepatitis C or Hepatitis B.
10. History of any other prior malignancy except for curatively treated basal cell or squamous cell carcinoma of skin, in situ cervical cancer, in situ breast cancer, in situ prostate cancer or any other cancer for which the subject has been diseasefree for at least 3 years.
11. Women who are pregnant or lactating.
12. Women of childbearing potential [defined as a sexually mature woman who has not undergone hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e. who has had menses any time in the preceding 24 consecutive months)] and men, not agreeing to use adequate contraception (e.g., hormonal or barrier method of birth control or abstinence) prior to study entry (after signing the informed consent document), during the duration of study participation and for at least 4 weeks after withdrawal from the study, unless they are surgically sterilised.
13. Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at an unacceptable risk or deems the subject not suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of P1446A-05 in subjects with advanced refractory malignancies | End of cycle 1 (3 weeks)

SECONDARY OUTCOMES:
1 To evaluate safety and tolerability ,pharmacokinetics of P1446A-05 in study population 2. To evaluate efficacy of P1446A-05 3. To perform exploratory analysis of biomarkers associated with use of P1446A-05 in the study population | End of cycle 1 (3 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Minish Jain, M.D., Principal Investigator — Consultant; Naresh Somani, D.M., Principal Investigator — Sr. Hemato-Oncologist & Pediatric Oncologist; Anish Maru, D.M., Principal Investigator — Senior Consultant and Director; Shona Nag, M.D., Principal Investigator — Consultant Medical Oncologist; Sudeep Gupta, D.M., Principal Investigator — Oncology Associate Professor
Locations (5):
- India (5):
  - Tata Memorial Centre, Mumbai, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Jehangir Hospital, Pune, Maharashtra
  - SEAROC Cancer Centre,, Jaipur, Rajasthan
  - Bhagwan Mahaveer Cancer Hospital, Jaipur, Rajasthan